CLINICAL TRIAL: NCT03959020
Title: Applying Long-term Follow-up to Improve Patient Selection in Laparoscopic Anti-reflux Surgery
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Sygehus Lillebaelt (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Jonas Sanberg Jensen, Ph.d.-student, University of Southern Denmark
Other Study IDs: JSJ_OP401
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: GERD; Reflux, Gastroesophageal; Surgery
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients, undergoing anti-reflux surgery: Patients having undergone anti-reflux surgery at the Department of Surgery, Kolding Hospital, a part of Hospital Lillebaelt, from 1th January 2002 - 31th December 2013
  Interventions: Procedure: Anti-reflux surgery

INTERVENTIONS:
Procedure: Anti-reflux surgery — Anti-reflux surgery for verified GERD

SUMMARY:
Introduction Laparoscopic anti-reflux surgery is considered standard of care in surgical treatment of gastro-oesophageal reflux disease and is not without risks of adverse effects, most notably disruption of the fundoplication, post-fundoplication dysphagia and gas-bloat-syndrome, in some cases leading to reoperation. Non-surgical factors such as pre-existing anxiety or depression disorders can influence postoperative satisfaction and symptom relief. Previous studies have focused on short-term follow-up or only certain aspects of disease, resulting in a less than complete picture.

The aim of this study is to evaluate long-term patient-satisfaction and durability of laparoscopic anti-reflux surgery in a large Danish cohort using comprehensive multimodal follow-up, and using the results of follow-up, to develop a clinically applicable scoring system usable in selecting patients for anti-reflux surgery.

Methods and analysis The study is a retrospective cohort study utilizing data from patient records and follow-up with patient-reported quality of life as well as registry-based data. The study population consists of all adult patients having undergone laparoscopic anti-reflux surgery at The Department of Surgery, Kolding Hospital, a part of Lillebaelt Hospital Denmark in an 11-year period. From electronic records; patient characteristics, preoperative endoscopic findings, reflux disease characteristics and details on type of surgery, will be identified. Disease specific quality-of-life and dysphagia will be identified from patient-reported follow-up. From Danish national registries, data on comorbidity, reoperative surgery, use of pharmacological anti-reflux treatment, mortality and socioeconomic factors will be included. Primary outcome of this study is treatment success at follow-up.

Ethics and dissemination For the study approval will be sought from The Danish Patient Safety Agency, The Danish Health Data Authority and Statistics Denmark, complying to Danish and EU current legislation. Inclusion in the study will require informed consent from participating subjects.

DETAILED DESCRIPTION:
Aim To use registry-based data and long-term quality of life follow up after anti-reflux surgery to quantify efficacy of treatment and to propose a clinically applicable tool to improve patient selection for surgery.

Background Treatment of GERD consists of anti-secretory drugs, mainly proton pump inhibitors, or anti-reflux surgery. Laparoscopic anti-reflux surgery is considered standard of care in surgical treatment of gastro-esophageal reflux disease and with careful patient selection based on thorough preoperative workup; symptom control and patient satisfaction are high compared to medical therapy).

Despite a tailored approach, laparoscopic anti-reflux surgery is not without risks of adverse effects, most notably disruption of the fundoplication, post-fundoplication dysphagia and gas-bloat-syndrome, in some cases leading to reoperation. Furthermore non-surgical factors such as pre-existing anxiety or depression disorders can influence postoperative satisfaction and symptom relief when compared to patients without concomitant psychological disorders.

Although few studies conclude that medical and surgical treatment of GERD have similar effectiveness, disease-specific quality of life generally improves after anti-reflux surgery and patient satisfaction is high. Depending on surgical procedure, the postoperative quality of life, ranges from significantly increased compared to preoperative measurements, to "normal" values as found in subjects devoid of GERD. 73-98% are satisfied with their condition after surgery and would choose surgery again.

Follow-up of randomized clinical trials have demonstrated, that anti-reflux surgery patients use acid suppressing drugs, primarily proton pump inhibitor (PPI) therapy at postoperative follow-up. Use have been considered minimal with <20% using PPI-therapy and 27-44% using PPI at five-year follow-up. A recent register-based study, demonstrated a greater number of redeemed prescriptions of proton pump inhibitor after primary anti-reflux surgery, than previously known. Five-, 10- and 15-year risks of long-term PPI use were 29.4%, 41.1% and 56.6%. However, this register-based study could not examine whether patients had objective recurrence of reflux disease and also did not examine indication for treatment as well as prescribing physician. From 2001 to 2011, 94,4% of PPI where prescribed in primary care and it is unknown why post-fundoplication patients are prescribed PPI. It has previously been demonstrated, that the use of acid suppressing drugs after anti-reflux surgery does not necessarily correlate with abnormal acid exposure to the esophagus . In general, the use of PPI has increased rapidly in Denmark, rising 243% from 2001 to 2011 despite more restrictive guidelines and changes in reimbursement . It must also be taken under consideration that although PPIs are a safe group of drugs, there are possible side effects such as increased risk of fractures, interaction with platelet inhibitor Clopidogrel, increased risk of kidney failure, pneumonia and hypomagnesaemia. As the majority of proton pump inhibitors are prescribed by general practitioners and not by the surgical centers, surgeons have very little knowledge of this aspect of life following anti-reflux surgery.

Laparoscopic anti-reflux surgery is more effective than medical management with regard to short to medium length follow-up. Few studies provide long-term follow-up. After ten years, the benefits of surgery seem to decrease, but there is still a significant improvement in quality of life compared to preoperative measurements . Known causes of dissatisfaction are postoperative complication, redo-fundoplication and developing new bothersome symptoms such as gas-bloat and dysphagia combined with inadequate symptom relief.

Hypothesis Long-term follow-up of anti-reflux surgery in combination with preoperative evaluation can be used to evaluate treatment success for a large cohort of patients and to create a clinically applicable tool for selecting patients for anti-reflux surgery predicting success of treatment.

Methods and materials Included in the study will be patients in the period 2002-2013 that had anti-reflux surgery at Department of Surgery, Kolding Hospital (n=557). Primary indication for surgery must be GERD (Nomesco: KJBC00-02).

Using patient records preoperative evaluation, including comorbidity and perioperative data will be registered. Postoperative complications within 30 days will be evaluated. Data on redo-surgery will be extracted from the National Patient Registry. 30-day mortality (National Civic Registry), data on socioeconomic status at primary surgery (The Integrated Database for Labour Market), preoperative use of PPI 2 years before primary surgery (Danish National Prescription Register) and information on psychiatric comorbidity (The Danish Psychiatric Central Research Register) will be extracted. All patients in the cohort will be contacted and included in follow-up evaluating specific quality of life (GERD-HRQL(59)) as well as dysphagia. They will also be asked whether they use any acid suppressing drugs, which physician prescribed them and the primary reason for use.

Statistical analysis Multiple logistic regression will be performed and used to establish significant preoperative and perioperative predictors for success of treatment. Failure of surgical treatment will be defined as any redo-surgery, consistent use of PPI postoperatively, significantly reduced quality of life or low patient satisfaction. Variables considered will be: demographics (age, sex, smoking, body mass index, employment status, educational level and income), endoscopic findings (esophagitis, hiatal hernia), symptoms of reflux (typical/atypical), comorbidity (ASA, Charlson Index, psychiatric comorbidity, previous abdominal surgery), pH-measurement (acid/non-acid reflux), esophageal manometry (normal, hyper- or hypomotility), preoperative quality of life and preoperative PPI-consumption as well as operative data (duration of surgery, length of stay, type of fundoplication, postoperative complications) respectively. Patients in the cohort having redo-surgery performed at any point since primary surgery will be selected for separate analysis examining comparing quality of life, patient satisfaction and predictive factors for redo-surgery. Survival analysis of fundoplication clinical durability will also be performed. The results will be used to create a clinically applicable scoring system facilitating successful preoperative evaluation before anti-reflux surgery.

Assuming 90% follow-up rate in the entire cohort, 501 patients will be included in the cohort. Retrospective data are available for all 557 patients. Reoperation, use of PPI and mortality will be extracted from registries yielding 100% follow-up under the assumption that no patient emigrated since surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone any anti-reflux surgery at Department of Surgery, Kolding Hospital, a part of Hospital Lillebaelt, Denmark from January 1, 2002 to December 31, 2013

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all adult patients (age +18) having undergone laparoscopic anti-reflux surgery (Nomesco Classification of Surgical Procedures (NCSP): KJBC01) from January 1, 2002 to December 31, 2013 in The Department of Surgery, Kolding Hospital, a part of Hospital Lillebaelt Denmark (n=557). Patients will be identified through Lillebaelt Hospital's Patient Administrative System. Day of surgery will be considered index date.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Treatment failure | From surgery to 1th January 2019 (Up to 17 years)
  Failure of anti-reflux surgery defined as
  1. Having undergone reoperation (NSCP: KJBC00-02, KJBW96-98, KJBB00-01, KJBB96-97) between index date and end of follow-up.
  2. Having filled prescription of >60 DDD/year of PPI in any year between index date and end of follow-up.
  3. Having no measure >3 on GERD-HRQL indicating symptoms being bothersome every day.
  4. Having no measure >4 on Dysphagia Handicap index indicating symptoms being a moderate problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Kolding Hospital, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanberg Ljungdalh J, Rubin KH, Durup J, Houlind KC. Long-term patient satisfaction and durability of laparoscopic anti-reflux surgery in a large Danish cohort: study protocol for a retrospective cohort study with development of a novel scoring system for patient selection. BMJ Open. 2020 Mar 16;10(3):e034257. doi: 10.1136/bmjopen-2019-034257. PMID 32184312

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03959020/Prot_SAP_000.pdf